CLINICAL TRIAL: NCT01914211
Title: The Role of Tranexamic Acid in Reducing Blood Transfusion Requirements After Cardiopulmonary Bypass in Neonates
Status: Withdrawn | Type: Observational
Sponsor: Aymen N Naguib (Other)
Responsible Party: Sponsor-Investigator, Aymen N Naguib, Director of Pediatric Cardiothoracic Anesthesia, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00350
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute Normovolemic Hemodilution: Patients that receive acute normovolemic hemodilution prior to surgery.
  Interventions: Procedure: Acute Normovolemic Hemodilution
- Tranexamic Acid: Patients that receive tranexamic acid during surgery.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 100mg/kg prior to incision, 100mg/kg on CPB and 100mg/kg after reversal of heparin with protamine.
  Groups: Tranexamic Acid
Procedure: Acute Normovolemic Hemodilution — Draw 20 mL/kg (up to 5Kg) of blood from patient and replace with washed PRBCs at 10-20mL/kg. (If > 5Kg draw 20% of circulating blood volume without PRBC replacement)
  Groups: Acute Normovolemic Hemodilution

SUMMARY:
This is an observational, prospective study to evaluate the role of tranexamic acid in reducing blood transfusion in neonates undergoing cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* All neonates undergoing arterial switch or aortic arch procedure utilizing cardiopulmonary bypass (CPB).

Exclusion Criteria:

* Jehovah's witness patients.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients from the cardiothoracic surgery population at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Level of postoperative hemostasis | 24 hours
  Evaluating the body's ability to stop or decrease postoperative bleeding.

SECONDARY OUTCOMES:
Volume of blood transfusions | 24 hours
  Assessing the need for and amount of blood transfusions during the 1st 24 hours post-op.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States